CLINICAL TRIAL: NCT04516044
Title: Long-term Followup of Effects of Customized Videogames on Physician Triage Practices
Brief Title: Effect of Videogames on Real-life Triage Patterns
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Deepika Mohan, Associate Professor of Critical Care Medicine, University of Pittsburgh
Other Study IDs: STUDY20070012; DP2LM012339 (NIH)
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Trauma; Physician's Role
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Video game: Patients treated by physicians who were randomized to either play an adventure-based video game that used narrative engagement to recalibrate physician heuristics in trauma triage or a puzzle-based video game that used analogical encoding to recalibrate physician heuristics in trauma triage.
  Interventions: Behavioral: Video games
- Control: Patients treated by physicians who were randomized either to nothing at all or to a text-based educational program.

INTERVENTIONS:
Behavioral: Video games — See arm description
  Groups: Video game

SUMMARY:
In 2016 and 2017 the investigators conducted two clinical trials in which emergency medicine physicians were randomized either to an intervention (customized, theoretically-based video games) or to a control (nothing or text-based education). This study will now assess long-term outcomes for physicians enrolled in those two trials to evaluate the effect of the interventions on triage practices for trauma patients who presented initially to non-trauma centers in the US between December 2016 and November 2018.

ELIGIBILITY:
Inclusion Criteria:

* Participated in two prior clinical trials (Physician)
* ≥65 years old (Patient)
* enrolled in Medicare fee-for-service
* sustained a moderate-severe injury (i.e. ISS [injury severity score] >15) (Patient)
* treated by physician enrolled in prior clinical trials (Patient)

Exclusion Criteria:

* Did not participate in two prior clinical trials (Physician)
* <65 years old (Patient)

Ages: 25 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 65 who presented after a moderate-severe injury to a non-trauma center in the US during 2016-2018.
Sampling Method: Non-Probability Sample
Enrollment: 686 (Actual)
Dates: Start 2016-10-30 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Number of patients triaged to trauma centers | 1 year following the intervention
  The investigators will use Medicare claims to measure the number of patients, treated by study participants, who present initially to non-trauma centers after a moderate-severe injury and are transferred to a Level I/II trauma center during that episode of care. They will compare triage patterns for patients treated by physicians in the intervention and in the control groups.

SECONDARY OUTCOMES:
Number of moderate-severely injured patients who die 30-days after initial evaluation | 1 year following the intervention
  Patient mortality 30-days after evaluation for a moderate-severe injury by a physician enrolled in the trial, compared among intervention and control groups.
Frequency of resources used for patients with moderate-severe injuries treated by participants | 1 year following intervention
  Frequency of resources used (e.g. ICU admission, mechanical ventilation, disposition status) after initial presentation for a moderate-severe injury and treatment by a participating physician, compared among intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Mohan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data is available for sharing, conditional on approval by the University of Pittsburgh Office of Research and Institutional Review Board.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 3 years
Access Criteria: Contact the PI

REFERENCES:
- [Background] Mohan D, Farris C, Fischhoff B, Rosengart MR, Angus DC, Yealy DM, Wallace DJ, Barnato AE. Efficacy of educational video game versus traditional educational apps at improving physician decision making in trauma triage: randomized controlled trial. BMJ. 2017 Dec 12;359:j5416. doi: 10.1136/bmj.j5416. PMID 29233854
- [Background] Mohan D, Fischhoff B, Angus DC, Rosengart MR, Wallace DJ, Yealy DM, Farris C, Chang CH, Kerti S, Barnato AE. Serious games may improve physician heuristics in trauma triage. Proc Natl Acad Sci U S A. 2018 Sep 11;115(37):9204-9209. doi: 10.1073/pnas.1805450115. Epub 2018 Aug 27. PMID 30150397